CLINICAL TRIAL: NCT04266561
Title: Laparoscopic Management of Recurrent Inguinal Hernia in Children
Brief Title: Laparoscopic Recurrent Inguinal Hernia Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Rafik Shalaby, Professor, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-30121949; Rafik-2015 (Registry Identifier: Al-Azhar University)
Record Dates: First submitted 2014-06-24; First posted 2020-02-12 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Congenital Hernia
Keywords: Laparoscopy; Recurrent inguinal hernia; Children
MeSH Terms: conditions — Hernia, Inguinal | interventions — Herniorrhaphy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lap. recurent inguinal hernia repair (Other): After induction of general anesthesia, the patient was placed supine in Trendelenburg's position. Insertion of the main umbilical port. Laparoscopic hernia repair was done by intracorporeal insertion of purse string technique with some modifications
  Interventions: Other: hernia repair

INTERVENTIONS:
Other: hernia repair — Two 3-mm needle holders were used for stitching the wide IIR. Then the suture was continued along the upper margin of IIR, but in a deeper plane to include the peritoneum and the deeper fascia transversalis.

SUMMARY:
Laparoscopic management of recurrent inguinal hernia in children has been recently introduced in surgical practice. One of the most important advantages of using the laparoscopic approach in cases with recurrent inguinal hernia (RIH) is that it avoids the previous operation site thus avoiding injuries to the vas and vessels [19]. Some authors designed a study to compare laparoscopic hernia repairs with classical open repairs for pediatric RIH following the ﬁrst open repair. They stated that avoiding the scarred tissue the former operation area with the laparoscopic approach facilitates the procedure and decreases both the operative time and complication rate. [5]. Further, it is as simple as a fresh hernia repair because the time taken for the repair of recurrent hernia laparoscopically was the same as the fresh laparoscopic repair with no added complication [5,20]. In laparoscopic surgery, approaching the hernia defect from within the abdomen, makes the area of interest bloodless, and the magnification renders anatomy very clear, making surgery precise [6,7].

DETAILED DESCRIPTION:
Abstract: Background: Open repair of recurrent inguinal hernias [RIH] in infancy and childhood is difficult and there is definite risk of damaging the vas deferens and testicular vessels. Laparoscopic repair of RIH has the benefit of avoiding the previous operative site. The aim of this study is to present the investigator's experience with laparoscopic repair of RIH either after open or laparoscopic hernia repair with stress on technical refinements to prevent recurrence. Patients and methods: This is a retrospective study of laparoscopic repair of recurrent inguinal hernia. Records of patients that have been subjected to laparoscopic inguinal hernia repair for RIH were reviewed and evaluated. All patients were subjected to laparoscopic repair of 42 recurrent hernial defects. The primary outcome measurements of this study include; operative time. The secondary outcomes include; hydrocele formation, iatrogenic ascent of the testis and testicular atrophy.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent inguinal hernia

Exclusion Criteria:

* complicated inguinal hernia

Ages: 6 Months to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2010-02; Primary Completion 2013-03 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Operative time | From the incision time to the closure of the wound
  The operative time is estimated by minutes. The estimated operative time for unilateral and bilateral recurrent hernia are estimated

SECONDARY OUTCOMES:
Hydrocele formation | one month postoperatively
  Clinical and ultrasound examination of the scrotum. Hydrocele is diagnosed by the presence of fluids in the tunica albugenia around the testis. It is measured by ml liter
Testicular atrophy | three months postoperatively
  Clinical and ultrasound examination of the testis for estimation of testicular size in cm.

CONTACTS AND LOCATIONS:
Overall Officials: Rafik Shalaby, MD, Principal Investigator — Al-Azhar University, Nasr City, Cairo, Egypt
Locations (1):
- Al-Housain University Hospital, Cairo, Egypt

REFERENCES:
- [Background] Shalaby R, Ismail M, Dorgham A, Hefny K, Alsaied G, Gabr K, Abdelaziz M. Laparoscopic hernia repair in infancy and childhood: evaluation of 2 different techniques. J Pediatr Surg. 2010 Nov;45(11):2210-6. doi: 10.1016/j.jpedsurg.2010.07.004. PMID 21034946
- [Background] Shalaby RY, Fawy M, Soliman SM, Dorgham A. A new simplified technique for needlescopic inguinal herniorrhaphy in children. J Pediatr Surg. 2006 Apr;41(4):863-7. doi: 10.1016/j.jpedsurg.2005.12.042. PMID 16567212
- [Background] Shalaby R, Ibrahem R, Shahin M, Yehya A, Abdalrazek M, Alsayaad I, Shouker MA. Laparoscopic Hernia Repair versus Open Herniotomy in Children: A Controlled Randomized Study. Minim Invasive Surg. 2012;2012:484135. doi: 10.1155/2012/484135. Epub 2012 Dec 27. PMID 23326656
- [Background] Shalaby R, Desoky A. Needlescopic inguinal hernia repair in children. Pediatr Surg Int. 2002 Mar;18(2-3):153-6. doi: 10.1007/s003830100655. PMID 11956783